CLINICAL TRIAL: NCT03546959
Title: Dynamic Lycra Orthosis as an Adjunct to Botulinum Toxin-A Injection of the Upper Limb in Adults Following Stroke: A Single-blinded Randomized Controlled Trial
Brief Title: Dynamic Lycra Orthosis as an Adjunct to Botulinum Toxin-A Injection for Post-stroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2017.677
Record Dates: First submitted 2018-05-12; First posted 2018-06-06 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2018-06

CONDITIONS: Stroke; Spasticity as Sequela of Stroke; Upper Limb Hypertonia
Keywords: stroke; spasticity; lycra; orthosis; splint; treatment; upper extremity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Rehabilitation; Botulinum Toxins

STUDY DESIGN:
Intervention Model Description: Paralel group randomized controlled study
Who Masked: Investigator, Outcomes Assessor
Masking Description: outcome assessor blinded to participants' allocated group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lycra sleeve after botulinum toxin (Experimental): 8 hours a day lycra sleeve wear plus rehabilitation (for five days a week for three weeks) after botulinum toxin injection for post-stroke spasticity
  Interventions: Other: Lycra sleeve; Other: Rehabilitation; Drug: Botulinum Toxin
- Rehabilitation after botulinum toxin (Active Comparator): Rehabilitation (five days a week for three weeks) after botulinum toxin injection for post-stroke spasticity
  Interventions: Other: Rehabilitation; Drug: Botulinum Toxin

INTERVENTIONS:
Other: Lycra sleeve — custom-fitted lycra sleeve extending from axilla to wrist
  Other Names: Rehabilitation after botulinum toxin injection
  Arms: Lycra sleeve after botulinum toxin
Other: Rehabilitation — Passive, active and active assistive range of motion and stretching exercises for shoulder, elbow, wrist, facilitation and inhibition techniques, neuromuscular electrical stimulation for wrist extensors, strengthening exercises for affected upper extremity, occupational therapy
  Other Names: botulinum toxin injection for post stroke spasticity
Drug: Botulinum Toxin — Botulinum toxin injection for upper limb spasticity after stroke
  Other Names: botulinum toxin injection for post stroke spasticity

SUMMARY:
Upper extremity splints are one of the nonpharmacologic treatments used to treat hypertonicity after stroke. The purpose of splinting is to support, to position, to immobilize, to prevent contracture and deformities, to reduce spasticity and to enhance function. Dynamic lycra splints have been found to improve spasticity, posture, and fluency of upper extremity movements in computerized analysis systems due to the effects of neutral warmth, circumferential pressure and by creating a low intensity prolonged stretch on hypertonic muscles , all of which contribute to increased sensory awareness of the involved limb. These splints are frequently used in the field of neurological rehabilitation, but there is not enough scientific evidence about their efficacy. It was demonstrated that lycra sleeves have positive effects on upper extremity function of children with cerebral palsy. Lycra sleeves for upper extremity function after stroke is a relatively new field of research.

The aim of this study is to investigate effects of dynamic lycra orthosis as an adjunct to botulinum toxin-a injection of the upper limb in adults following stroke.

DETAILED DESCRIPTION:
Spasticity is defined as a velocity-dependent increase in muscle tone resulting from hyper-excitability of the tonic stretch reflex in people with upper motor neurone (UMN) syndrome following damage to the brain or spinal cord. If left untreated, a vicious cycle occurs, in which unopposed contraction (spastic dystonia) in the affected muscle groups leads to an abnormal limb posture, resulting in soft tissue shortening and further biomechanical changes in the contracted muscles. This in turn prevents muscle lengthening and further stiffness. Botulinum toxin type A (BoNT-A) has been shown to provide a sustained reduction in post-stroke upper-limb spasticity when combined with rehabilitation. Although the trial-based evidence for enhanced benefit through a combination of BoNT-A and physical intervention is limited, the benefits of a combined approach are well-accepted in clinical practice. A successful treatment package, often incorporating physical and pharmacological treatments, can improve physical function and can also prevent secondary complications. A recent systematic review concluded that there is an urgent need for large-scale, rigorous clinical trials that investigate the relative efficacy of therapy types as independent or combined interventions with BoNT-A injection.

Dynamic lycra splints are proposed to modify hypertonicity due to the effects of neutral warmth, circumferential pressure and by creating a low intensity prolonged stretch on hypertonic muscles, all of which contribute to increased sensory awareness of the involved limb. Lycra arm splints comprise circumferential lycra segments that are orientated to produce a specific 'direction of pull'. Lycra1 arm splints specifically aim to influence hypertonicity, posture and patterns of movement. All of which are expected to result in improved movement performance, particularly fluency or smoothness of movement and to contribute to improved function. It was demonstrated that lycra sleeves have positive effects on upper extremity function of children with cerebral palsy. Lycra sleeves for upper extremity function after stroke is a relatively new field of research. The aim of this study is to investigate effects of dynamic lycra orthosis as an adjunct to botulinum toxin-a injection of the upper limb in adults following stroke.

Patients with stroke for more than three months and who are in need for botulinum toxin injection for post-stroke upper limb spasticity will be randomized to two groups: Lycra sleeve plus rehabilitation and only rehabilitation groups. After botulinum toxin injection, both groups will receive rehabilitation program including passive, active and active assistive range of motion and stretching exercises for shoulder, elbow, wrist, facilitation and inhibition techniques, neuromuscular electrical stimulation for wrist extensors, strengthening exercises for affected upper extremity, occupational therapy for two hours a day, five days a week for three weeks. Intervention group will wear lycra sleeve for eight hours a day, five days a week for three weeks. Effects of lycra sleeves as an adjunct to rehabilitation program after botulinum toxin injection will be assessed by using Fugl Meyer Upper Limb Motor score and Motricity index for motor function, Modified Ashworth scale for spasticity, Box and Block test score for hand dexterity, Semmes-Weinstein monofilaments for sensory functions. Outcome assessment will be undertaken by a blinded assessor at before treatment, after treatment (at 3 weeks) and after three months.

Friedman test will be used to establish within group changes over time in outcome variables. Wilcoxon's signed-rank test will be performed to show differences in the parameters between baseline and follow-up points. Between groups differences will be analyzed by using Mann-Whitney U test. Results will be considered significant when P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Adult stroke (18-80 years)
2. Patients with stroke who can sit without support
3. Patients with stroke who have spasticity which limit upper limb function

Exclusion Criteria:

1. Brunnstrom motor recovery stage 1 and 6
2. Comorbidities such as hemiplegic shoulder pain, complex regional pain syndrome, central post-stroke pain, brachial plexus injury etc.
3. Upper limb spasticity with MAS level 4 or presence of contracture in upper extremity.
4. Contraindications for lycra sleeve ( circulatory disorder etc.)
5. Contraindications for botulinum toxin (infection at the injection site, hypersensitivity to toxin etc.)
6. Severe aphasia or cognitive dysfunction that limit participation in rehabilitation (7) Receiving botulinum toxin injection within the last 6 months

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Motor Assessment Scale | Day 0
  Fugl-Meyer Upper Extremity Assessment assesses motor impairment in the upper extremities. There is no total score for this measure. Sub-scales include: upper extremity (0-36), wrist (0-10), hand (0-14), coordination/speed (0-6) (which can be combined to form a total motor function score out of 66). Higher scores indicate better performance.
Fugl-Meyer Upper Extremity Motor Assessment Scale | 3 weeks
  Fugl-Meyer Upper Extremity Assessment assesses motor impairment in the upper extremities. There is no total score for this measure. Sub-scales include: upper extremity (0-36), wrist (0-10), hand (0-14), coordination/speed (0-6) (which can be combined to form a total motor function score out of 66). Higher scores indicate better performance.
Fugl-Meyer Upper Extremity Motor Assessment Scale | 3 months
  Fugl-Meyer Upper Extremity Assessment assesses motor impairment in the upper extremities. There is no total score for this measure. Sub-scales include: upper extremity (0-36), wrist (0-10), hand (0-14), coordination/speed (0-6) (which can be combined to form a total motor function score out of 66). Higher scores indicate better performance.

SECONDARY OUTCOMES:
Motricity Index Upper Limb | Day 0
  Upper limb motor function Resistance to pinch, elbow flexion and shoulder abduction are scored to a maximum score of 33. Section scores are summed to a total of 100.
  0 = No movement.
  9 = Palpable contraction in muscle but no movement.
  14 = Movement seen but not full range/ not against gravity.
  19 = Full range against gravity, not against resistance.
  25 = Movement against resistance but weaker than other side.
  33 = Normal power.
Motricity Index Upper Limb | 3 weeks
  Upper limb motor function Resistance to pinch, elbow flexion and shoulder abduction are scored to a maximum score of 33. Section scores are summed to a total of 100.
  0 = No movement.
  9 = Palpable contraction in muscle but no movement.
  14 = Movement seen but not full range/ not against gravity.
  19 = Full range against gravity, not against resistance.
  25 = Movement against resistance but weaker than other side.
  33 = Normal power.
Motricity Index Upper Limb | 3 months
  Upper limb motor function Resistance to pinch, elbow flexion and shoulder abduction are scored to a maximum score of 33. Section scores are summed to a total of 100.
  0 = No movement.
  9 = Palpable contraction in muscle but no movement.
  14 = Movement seen but not full range/ not against gravity.
  19 = Full range against gravity, not against resistance.
  25 = Movement against resistance but weaker than other side.
  33 = Normal power.
Box and Block Test (BBT) | Day 0
  Evaluates gross manuel dexterity. Box and Block Test which consists of a box divided into two compartments by a partition and blocks with standardized dimensions is used to assess unilateral gross manuel dexterity. The object is instructed to transport boxes one by one from one compartment of the box to other in 60 seconds. The object should sit on a chair with a standard height and face the box. He/she should practice for a 15 second trial period before testing. If two blocks are carried at the same time, it is counted as one. And also if the block falls on the floor after it has been carried across, it is still counted. The score is the number of boxes transferred from one compartment to other in 60 seconds.
Box and Block Test (BBT) | 3 weeks
  Evaluates gross manuel dexterity. Box and Block Test which consists of a box divided into two compartments by a partition and blocks with standardized dimensions is used to assess unilateral gross manuel dexterity. The object is instructed to transport boxes one by one from one compartment of the box to other in 60 seconds. The object should sit on a chair with a standard height and face the box. He/she should practice for a 15 second trial period before testing. If two blocks are carried at the same time, it is counted as one. And also if the block falls on the floor after it has been carried across, it is still counted. The score is the number of boxes transferred from one compartment to other in 60 seconds.
Box and Block Test (BBT) | 3 months
  Evaluates gross manuel dexterity. Box and Block Test which consists of a box divided into two compartments by a partition and blocks with standardized dimensions is used to assess unilateral gross manuel dexterity. The object is instructed to transport boxes one by one from one compartment of the box to other in 60 seconds. The object should sit on a chair with a standard height and face the box. He/she should practice for a 15 second trial period before testing. If two blocks are carried at the same time, it is counted as one. And also if the block falls on the floor after it has been carried across, it is still counted. The score is the number of boxes transferred from one compartment to other in 60 seconds.
Semmes-Weinstein monofilaments for sensory functions digit 1 | Day 0
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 2 | Day 0
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 4 | Day 0
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 5 | Day 0
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 1 | 3 weeks
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 2 | 3 weeks
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 4 | 3 weeks
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 5 | 3 weeks
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 1 | 3 months
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 2 | 3 months
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 4 | 3 months
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Semmes-Weinstein monofilaments for sensory functions digit 5 | 3 months
  Assess touch detection thresholds of the fingers. 5 filaments from 0.07 gram to 279 grams will be used. Five different positions of the hand are tested: fingertip on digit 1,2,4 and 5.
Modified Ashworth Scale (MAS) of elbow flexor | Day 0
  elbow flexor muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion (ROM) 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale (MAS) of wrist flexor | Day 0
  wrist flexor muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale (MAS) of elbow flexor | 3 weeks
  elbow flexor muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale (MAS) of wrist flexor | 3 weeks
  wrist flexor muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale (MAS) of elbow flexor | 3 months
  elbow flexor muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale (MAS) of wrist flexor | 3 months
  wrist flexor muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Stroke Impact Scale Version 3.0 (SIS 3.0) | Day 0
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life. It contains 59 items measuring 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week.
Stroke Impact Scale Version 3.0 (SIS 3.0) | 3 weeks
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life. It contains 59 items measuring 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week.
Stroke Impact Scale Version 3.0 (SIS 3.0) | 3 months
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life. It contains 59 items measuring 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gunduz, Prof, Study Chair — Marmara University
Locations (1):
- Esra Giray, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gracies JM, Marosszeky JE, Renton R, Sandanam J, Gandevia SC, Burke D. Short-term effects of dynamic lycra splints on upper limb in hemiplegic patients. Arch Phys Med Rehabil. 2000 Dec;81(12):1547-55. doi: 10.1053/apmr.2000.16346. PMID 11128888
- [Background] Elliott C, Reid S, Hamer P, Alderson J, Elliott B. Lycra((R)) arm splints improve movement fluency in children with cerebral palsy. Gait Posture. 2011 Feb;33(2):214-9. doi: 10.1016/j.gaitpost.2010.11.008. Epub 2010 Dec 4. PMID 21131201
- [Background] Elliott CM, Reid SL, Alderson JA, Elliott BC. Lycra arm splints in conjunction with goal-directed training can improve movement in children with cerebral palsy. NeuroRehabilitation. 2011;28(1):47-54. doi: 10.3233/NRE-2011-0631. PMID 21335677
- [Background] Nicholson JH, Morton RE, Attfield S, Rennie D. Assessment of upper-limb function and movement in children with cerebral palsy wearing lycra garments. Dev Med Child Neurol. 2001 Jun;43(6):384-91. doi: 10.1017/s001216220100072x. PMID 11409827
- [Background] Gracies JM, Fitzpatrick R, Wilson L, Burke D, Gandevia SC. Lycra garments designed for patients with upper limb spasticity: mechanical effects in normal subjects. Arch Phys Med Rehabil. 1997 Oct;78(10):1066-71. doi: 10.1016/s0003-9993(97)90129-5. PMID 9339154
- [Derived] Giray E, Gencer Atalay K, Eren N, Gunduz OH, Karadag-Saygi E. Effects of dynamic lycra orthosis as an adjunct to rehabilitation after botulinum toxin-A injection of the upper-limb in adults following stroke: A single-blinded randomized controlled pilot study. Top Stroke Rehabil. 2020 Sep;27(6):473-481. doi: 10.1080/10749357.2019.1704371. Epub 2019 Dec 23. PMID 31868130